CLINICAL TRIAL: NCT00715260
Title: A Multicenter, Prospective, Observational Study of Pruritus Amongst Hemodialysis Patients: The ITCH National Registry
Brief Title: An Observational Study of Pruritus Amongst Hemodialysis Patients
Acronym: ITCH Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Acologix, Inc. (Industry)
Responsible Party: Dawn McGuire, M.D. Chief Medical Officer, Acologix, Inc.
Other Study IDs: AC120-8002
Record Dates: First submitted 2008-07-08; First posted 2008-07-15 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Pruritus; Kidney Failure, Chronic; Hemodialysis; Chronic Disease
MeSH Terms: conditions — Pruritus; Kidney Failure, Chronic; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- UP Patients on HD: Uremic Pruritus (UP) patients maintained on hemodialysis (HD)

SUMMARY:
The purpose of this observational study is to better understand the natural history/natural course of uremic pruritus (UP) - itching associated with chronic kidney disease(CKD). During the lifetime of a CKD dialysis patient, UP tends to be a prolonged, frequent, and an intense itch that is known to impair the patient's quality of life (QoL), including sleep and mood.

The study will follow hemodialysis (HD) patients longitudinally to characterize their pruritus over time. The study will quantify and characterize UP and assess change over time; collect data on conditions that may be affected by UP such as sleep, mood, socialization and overall quality of life; collect data on use of medications, particularly anti-pruritic treatments, sleep aids, and medications for depression and anxiety; and collect data on medical resource use, particularly hospitalizations for treatment of skin and other infections over the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years;
* Patients receiving chronic hemodialysis 3 or more times per week;
* Patients who have "mild", "moderate" or "severe" pruritus;

  * "Mild" pruritus is defined as a nighttime or daytime worst itch intensity VAS >10 mm and < 40 mm at Screening and a combined daytime and nighttime Kawashima Itch Severity Score of < 2;
  * "Moderate" pruritus is defined as a nighttime or daytime worst itch intensity VAS >10 mm and < 40 mm at Screening and a combined daytime and nighttime Kawashima Itch Severity Score of ≥ 3;
  * "Severe" pruritus is defined as a nighttime or daytime worst itch intensity VAS of ≥ 40 mm at Screening and a combined daytime and nighttime Kawashima Itch Severity Score of ≥ 3;
* Patients who are able to understand and complete questionnaires written in English;
* Patients who are expected to continue to dialyze at the present dialysis unit for the duration of the study.

Exclusion Criteria:

* Patients who have pruritus attributed to causes other than chronic kidney disease (CKD) or the direct consequences of CKD (i.e., hyperparathyroidism, circulating "uremic toxins");
* Patients who have had significant alteration in their dialysis regimen within the 2 weeks prior to Screening (or those for whom such changes are anticipated during the study) are excluded. A "significant alteration" is defined as:

  * A change in the type of hemodialysis filter;
  * An increase or decrease in total duration of dialysis prescribed of > 1 hour/week;
  * A change in the site or type of venous access for dialysis;
  * An increase or decrease in prescribed blood flow of >100 mL/min;
* Patients who are unwilling to comply with the study protocol. Test Product, Dose, Mode of Administration and Duration of Treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on thrice-weekly (or more frequent) maintenance hemodialysis who have Uremic Pruritus
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn McGuire, M.D., Study Director — Acologix, Inc.
Locations (5):
- United States (5):
  - Kidney Care Associates, Augusta, Georgia
  - FMC Metaire, Metaire, Louisiana
  - Western New England Renal Associates, Springfield, Massachusetts
  - Southeast Renal Associates, Charlotte, North Carolina
  - Nephrology Associates, Chattanooga, Tennessee